CLINICAL TRIAL: NCT06843265
Title: Outcomes and Perceptions of the Implementation of the JADA Device in a Stage II Postpartum Hemorrhage Management Protocol in Referral Hospitals of the Colombian Pacific Region: a Cohort Study
Brief Title: Outcomes and Perceptions of the Implementation of the JADA Device in a Stage II Postpartum Hemorrhage Management Protocol in Referral Hospitals of the Colombian Pacific Region
Acronym: JADAValle
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Fundacion Clinica Valle del Lili (Other)
Collaborators: Hospital Universitario del Valle Evaristo Garcia (Unknown)
Responsible Party: Principal Investigator, María Fernanda Escobar, Global health equity unit director, Fundacion Clinica Valle del Lili
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2024.271
Record Dates: First submitted 2025-02-14; First posted 2025-02-24 (Actual); Last update posted 2025-02-24 (Actual); Status verified 2025-02

CONDITIONS: Post Partum Haemorrhage
Keywords: maternal mortality; Shock Index; care bundle
MeSH Terms: conditions — Postpartum Hemorrhage; Maternal Death

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Group 1 (Experimental): Pregnant women with stage II postpartum hemorrhage, after vaginal delivery, who have had the JADA device implemented and meet INVIMA's definition of use of the instrument: the JADA system is intended to provide control and treatment of abnormal postpartum uterine bleeding or postpartum hemorrhage when conservative management is warranted, attended in hospitals in the context of the Godfather Hospital Strategy in the department of Valle del Cauca.
  Interventions: Device: Vacuum- Induce Hemorrhage Control

INTERVENTIONS:
Device: Vacuum- Induce Hemorrhage Control — The JADA System is designed for single use only and is composed of medical grade silicone. Its components include an intrauterine loop with protected vacuum pores, a cervical seal with a sealing valve for infusing saline and a vacuum connector port for applying suction. The intrauterine loop is located at the distal end of a tube and contains 20 protected vacuum pores oriented inward along the loop. This shielded design facilitates intracavitary suction by shielding maternal tissue from the vacuum source and prevents clogging of the vacuum pores with tissue or clot.

SUMMARY:
This study focuses on postpartum hemorrhage (PPH), a condition that stands out as the leading cause of global maternal mortality. Annually, about 14 million women experience PPH, resulting in approximately 70,000 deaths. This condition presents a higher risk in low- and middle-income countries (LMICs), particularly where access to quality care is limited. Recognizing the urgency of addressing this public health problem, the Colombian Ministry of Health and Social Protection has implemented the Maternal Mortality Reduction Acceleration Plan (PARE) to improve maternal mortality indicators and meet the Sustainable Development Goals (SDGs).

The project will evaluate the results and perception of a new device in the management of stage II PPH in referral hospitals in the department of Valle del Cauca, integrated in the Hospital Padrino strategy. This initiative seeks not only to improve the understanding and treatment of PPH, but also to strengthen institutional capacities through education, creation of telecare networks and care services adapted to local needs.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women who are admitted to the obstetrics service scheduled for vaginal delivery in any of the participating hospitals: Fundación Valle del Lili, Hospital Universitario del Valle and Hospital Luis Ablanque de la Plata.
* Patient admitted during the shift of one of the gynecologists trained in the use of the JADA device in the context of the research project.

Criteria for the use of JADA device:

* Pregnant women over or equal to 18 years of age.
* Gestational age of pregnancy greater than 32 weeks of gestation.
* Pregnant with vaginal delivery.
* Pregnant with postpartum hemorrhage due to uterine atony that does not respond to treatment with uterotonics and uterine massage.
* Postpartum hemorrhage uterine stage/stage II.
* Vaginal delivery attended in a health institution in the context of the Hospital Padrino strategy (Fundación Valle del Lili or Hospital Universitario del Valle or Hospital Luis Ablanque de la Plata).

Exclusion Criteria:

* Patients who, according to the attending physician's criteria, are not candidates for vaginal delivery.
* Abnormality of the normal uterine anatomy.
* Placental abnormalities.
* Maternal anemia with hemoglobin less than 7 mg/dl prior to delivery.
* Those who do not sign informed consent.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — women by birth
Enrollment: 24 (Estimated)
Dates: Start 2025-06-01 (Estimated); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Bleeding control | up to 42 days postpartum
  Postpartum hemorrhage defined as quantified bleeding of more than 500 ml for vaginal deliveries and more than 1000 ml for cesarean deliveries, occurring within the first 24 h after delivery and which may be associated with signs of hemodynamic instability, i.e. the ratio between heart rate and systolic blood pressure (shock index).
  Following this concept of the shock index and the amount of bleeding, the stages of postpartum hemorrhage are divided, which, according to the result of the shock index, the therapy is directed:
  Stage 1: Bleeding 500-1000 cc, Shock index of <0.9, bleeding time <10 minutes. Stage 2: Bleeding 1000-1500 cc, shock index 0.9-1.4 bleeding time 10-20 minutes.
  Stage 3: Bleeding <1500 cc, shock index >1.5, bleeding time greater than 20 minutes.
  Stage 4: Cardiovascular collapse with profound hypovolemic shock and coagulopathy.
  These stages will be measured through a bag which will fulfill the function of measuring to indicate the stage and amount of bleeding

IPD SHARING:
Plan to Share IPD: Undecided
If the Colombian regulations request it, then it would be made